CLINICAL TRIAL: NCT01739816
Title: Polymedication Check - Evaluation of the Impact of Community Pharmacy Based Medication Review on Medicines Use and Humanistic Outcomes
Brief Title: Polymedication Check - a Randomised Controlled Trial
Acronym: evalPMC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kurt Hersberger (Other)
Collaborators: University of Basel (Other); University Hospital, Basel, Switzerland (Other); Polyclinique Médicale Universitaire, PMU, Lausanne (Unknown); Swiss Pharmacy Association, pharmaSuisse (Unknown)
Responsible Party: Sponsor-Investigator, Kurt Hersberger, Professor, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: evalPMC
Record Dates: First submitted 2012-11-27; First posted 2012-12-04 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Polypharmacy
Keywords: Compliance; Adherence; Polypharmacy; Medicines use; Medication review; Pharmaceutical care; Primary care; Drug related problem; Patient safety
MeSH Terms: conditions — Patient Compliance | interventions — Medication Review

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control group (No Intervention): Patients get no intervention at study start, but only at study end after seven months.
- Intervention group (Active Comparator): At the beginning and at the end of the study, this group receives a pharmacist's led medication review focusing on daily medicines use (= Polymedication Check).
  Interventions: Behavioral: Medication review
- Observational arm (Other): If participants after recruitment violate inclusion criteria (e.g. change from autonomous medication management to external home care) or insists on intervention despite being randomised to control group or patient condition forces pharmacist to provide a PMC.
  Interventions: Behavioral: Medication review

INTERVENTIONS:
Behavioral: Medication review — Polymedication Check (PMC) is a pharmacist's led medication review focusing medicines management, adherence issues and other drug related problems.
  The PMC has been implemented in 2010 as a new cognitive service provided by any community pharmacist to patient with polypharmacy (n>3 drugs) on long term conditions (> months). This specialised medication review follows a structured predefined protocol and is reimbursed by swiss health insurances.
  As an outcome, pharmacist may install a compliance support e.g. weekly filled pill organizer.
  Other Names: Polymedication Check
  Arms: Intervention group; Observational arm

SUMMARY:
Since October 2010, Swiss community pharmacies can offer a 'Polymedication Check' (PMC) to patients on ≥4 prescribed drugs taken over ≥3 months.

Aims:

To evaluate first experiences shortly after implementation, missed pharmaceutical care issues and barriers to implementation on pharmacist's level as well as patient's acceptance through qualitative and descriptive studies To evaluate the impact of PMC in Swiss primary Care and to evaluate economic, clinical and humanistic outcomes in a subsequent randomized controlled trial.

DETAILED DESCRIPTION:
Evaluating the newly implemented Swiss 'Polymedication-Check', a specialised medication review and screening for adherence issues, offers a large field of interesting research questions. Using the current PMC-Protocol as a structured interview guide, pharmacists are able to document their counselling on medication use issues and other drug related problems.

In a randomized-controlled trial we aim at analysing 800 recruited patients from 70 study pharmacies during seven months. Patients were recruited in the regions Basel, Aargau-Solothurn, Waadt in Switzerland and randomised using 1:1 block randomisation.

Primary outcome focuses on the improvement of adherence and persistence after 'Polymedication Check' (using medication possession ratio (MPR), gaps in medicines history records and patient's interviews).

Second outcomes are time to planned or unplanned consulting with a physician or hospitalisation, knowledge, safety of medicines use and patients management of polypharmacy.

ELIGIBILITY:
Inclusion Criteria:

* more than 3 drugs over at least 3 months prior to recruitment
* german or french language (written and spoken)
* medicines use in self management

Exclusion Criteria:

* provision of Polymedication Check in the past
* living in a nursing home
* use of prefilled pill organiser or individually blistered medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2012-06; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Medication possession ratio (MPR), gaps and persistence in medicines use | Seven months after recruitment
  Improvement of adherence seven months after 'Polymedication-Check' using medication possession ratio (MPR), gaps and persistence out of history records from community pharmacy.

SECONDARY OUTCOMES:
Time to planned or unplanned consulting with a physician or hospitalisation | Seven months after recruitment
  Time to planned or unplanned consulting with a physician or hospitalisation
Patient knowledge about his medicines | After two weeks, four and seven months after recruitment
  Patient knowledge about his medicines use, assessed through PMC (intervention goup) and two telephone interviews (both groups)
Self reported adherence | At study start and two weeks, four and seven months after after recruitment
  Self report of adherence: is assessed with self administrated questionnaires and telephone interviews
Patients safety | After two weeks, four and seven months after recruitment
  Patients safety is assessed through a) telephone interview with a focus on perceived safety and b) number of drug related problems addressed and solved at study end.

OTHER OUTCOMES:
Use of compliance aids | At study start and two weeks, four and seven months after after recruitment
  Compliance aids may be in use prior to recruitment, recommended after intervention by pharmacist, recommendation can be refused or accepted and the compliance aid can be filled by the patient himself or specialised service from the pharmacy.

CONTACTS AND LOCATIONS:
Overall Officials: Kurt E Hersberger, Prof., Study Director — University of Basel; Markus Messerli, MSc, Principal Investigator — University of Basel
Locations (1):
- Pharmaceutical Care Research Group, University of Basel, Basel, Basel, Switzerland

REFERENCES:
- [Background] Vrijens B, De Geest S, Hughes DA, Przemyslaw K, Demonceau J, Ruppar T, Dobbels F, Fargher E, Morrison V, Lewek P, Matyjaszczyk M, Mshelia C, Clyne W, Aronson JK, Urquhart J; ABC Project Team. A new taxonomy for describing and defining adherence to medications. Br J Clin Pharmacol. 2012 May;73(5):691-705. doi: 10.1111/j.1365-2125.2012.04167.x. PMID 22486599
- [Background] Krska J, Avery AJ; Community Pharmacy Medicines Management Project Evaluation Team. Evaluation of medication reviews conducted by community pharmacists: a quantitative analysis of documented issues and recommendations. Br J Clin Pharmacol. 2008 Mar;65(3):386-96. doi: 10.1111/j.1365-2125.2007.03022.x. Epub 2007 Oct 8. PMID 17922887
- [Background] Clifford S, Barber N, Elliott R, Hartley E, Horne R. Patient-centred advice is effective in improving adherence to medicines. Pharm World Sci. 2006 Jun;28(3):165-70. doi: 10.1007/s11096-006-9026-6. Epub 2006 Sep 27. PMID 17004019
- [Background] Kwint HF, Faber A, Gussekloo J, Bouvy ML. Effects of medication review on drug-related problems in patients using automated drug-dispensing systems: a pragmatic randomized controlled study. Drugs Aging. 2011 Apr 1;28(4):305-14. doi: 10.2165/11586850-000000000-00000. PMID 21428465
- [Background] Bryant LJ, Coster G, Gamble GD, McCormick RN. The General Practitioner-Pharmacist Collaboration (GPPC) study: a randomised controlled trial of clinical medication reviews in community pharmacy. Int J Pharm Pract. 2011 Apr;19(2):94-105. doi: 10.1111/j.2042-7174.2010.00079.x. Epub 2011 Feb 25. PMID 21385240
- [Derived] Messerli M, Blozik E, Vriends N, Hersberger KE. Impact of a community pharmacist-led medication review on medicines use in patients on polypharmacy--a prospective randomised controlled trial. BMC Health Serv Res. 2016 Apr 23;16:145. doi: 10.1186/s12913-016-1384-8. PMID 27108410
- See also: For recent publications, see 'Publications' -> 'Publications' and 'Posters' — http://www.pharmacare.unibas.ch